CLINICAL TRIAL: NCT00951951
Title: Gait Analysis of Anterior vs. Posterior Approach in Performance of Total Hip Arthroplasty: A Multi-Centre, Prospective Trial
Brief Title: Gait Analysis of Anterior Versus Posterior Approach in Performance of Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta USA (Industry)
Collaborators: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0001
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterior Surgical Approach (Active Comparator): (AMIS)
  Interventions: Procedure: Anterior Approach
- Posterior Approach Group (Active Comparator): Posterior surgical approach for total hip replacement.
  Interventions: Procedure: Posterior Approach

INTERVENTIONS:
Procedure: Anterior Approach — Anterior Minimal Invasive Surgery (AMIS)
  Arms: Anterior Surgical Approach
Procedure: Posterior Approach
  Other Names: Posterior Surgical Approach
  Arms: Posterior Approach Group

SUMMARY:
The primary objectives of the study is to compare gait kinematics and the return to normalization of gait in patients that have undergone a Total Hip Arthroplasty (THA) via the direct anterior approach versus the posterior approach. Gait kinematics will be measured using the IDEEA LifeGait device from Minisun (Fresno, CA).

DETAILED DESCRIPTION:
This is a prospective study of two different surgical approaches to THA, direct anterior vs posterior approach in approximately 64 patients that meet the standard criteria for the implantation of primary total hip replacement utilizing the Medacta implants and have elected to undergo THA.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the standard criteria for the implantation of primary total hip arthroplasty
* Those presenting with primary or secondary osteoarthritis
* Those presenting with disease that meets the indications for use for Medacta USA implants defined by this study (on-label use)

Exclusion Criteria:

* Pregnant women or women who plan to conceive within the year following surgery
* Inflammatory arthritic condition
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems
* Those already treated with a failed Total Hip Arthroplasty (THA)
* Muscle contracture around the hip joint
* Individuals who have undergone organ transplant
* Those with a known co-existent medical condition where death is anticipated within five years due to the pre-existing medical condition.
* Those with one or more medical conditions identified as a contraindication defined by the labeling on any Medacta implants used in this study
* Individuals who have had a THA on the contra-lateral side within the 6 months.
* Individuals who have undergone a THR on the contra-lateral side and whose outcome is considered unsatisfactory or not good
* Individuals requiring bilateral hip replacement
* Individuals whose body mass index (BMI; kg/m2) >40
* Individuals with active or suspected infection or sepsis
* Individuals with chronic renal failure as defined by the need for dialysis
* Patients with severe forms of developmental dysplasia of the hip (DDH): Crowe types II, III, IV
* History of drug and/or substance abuse

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Compare gait kinematics and the return to normalization of gait in patients that have undergone a THA via the direct anterior approach vs. the posterior approach. | Pre-Op, (2 weeks if fully ambulatory), 6 weeks, 3 months, 1 year

SECONDARY OUTCOMES:
Evaluate/compare two surgical approaches (direct anterior vs. posterior): Patient improvement (subjective and objective) following THA using the HHS. Patient overall function and pain following THA using the WOMAC. Post operative radiological findings | Pre-Op, 6 weeks, 3 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Goldberg, MD, Study Director — Medacta USA Medical Director
Locations (4):
- United States (4):
  - Sun Valley Orthopedic Surgeons, Surprise, Arizona
  - D. Kevin Lester, MD, Fresno, California
  - Peak Orthopedics, Lone Tree, Colorado
  - Intermountain Healthcare, St. George, Utah

REFERENCES:
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/osteoarthritis.html